CLINICAL TRIAL: NCT01380678
Title: A Randomized Controlled Trial of Intralesional Bevacizumab Injection on Primary Pterygium: Preliminary Results
Brief Title: Intralesional Bevacizumab Injection on Primary Pterygium
Acronym: bevacizumab
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Olan Suwan-apichon, Department of Ophthalmology, Faculty of medicine, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KKU-1007
Record Dates: First submitted 2010-06-14; First posted 2011-06-27 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2010-07

CONDITIONS: Pterygium; Inflammation
Keywords: bevacizumab; pterygium; treatment; elevation
MeSH Terms: conditions — Pterygium; Inflammation | interventions — Bevacizumab; Histamine Antagonists; Vasoconstrictor Agents

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevacizumab (Active Comparator): intralesional bevacizumab injection
  Interventions: Drug: Intralesional injection of bevacizumab
- Topical antihistamine and vasoconstrictor (Active Comparator): combination of topical antazoline HCl 0.05% and tetrahydrozoline HCl 0.04%
  Interventions: Drug: Topical antihistamine and vasoconstrictor

INTERVENTIONS:
Drug: Intralesional injection of bevacizumab — single dose of 2 mg of bevacizumab intralesional injection on pterygium Combination of topical antazoline and tetrahydrozoline four times a day
  Other Names: Avastin
  Arms: bevacizumab
Drug: Topical antihistamine and vasoconstrictor — combination of topical antazoline HCl 0.05% and tetrahydrozoline HCl 0.04%
  Other Names: Hista-oph
  Arms: Topical antihistamine and vasoconstrictor

SUMMARY:
The purpose of this study is to evaluate that intralesional injection of bevacizumab on primary pterygium can reduce the corneal pterygium area, inflammation, redness and other symptoms.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of intralesional injection of bevacizumab on primary pterygium treatment

ELIGIBILITY:
Inclusion Criteria:

* primary pterygium

Exclusion Criteria:

* previous ocular surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
percentage of corneal pterygium area | 3 years
  Prior to receive the treatments, patients were asked to evaluate grading of their own symptoms and underwent clinical grading of the elevation and inflammation of the lesions using slit lamp biomicroscopy by an opthalmologist (OE). Digital photographs of each eye with pterygium were obtained for corneal pterygium area analysis [Sony Mavica digital still camera MVC-FD83, Japan]. Each patient was randomly assigned into either treatment group or control group using computer-generated random numbers table.
  Number of patients with adverse events will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Olan Suwan-apichon, md, Principal Investigator — Khon Kaen University
Locations (1):
- Srinagarind Hospital, Mueng, Changwat Khon Kaen, Thailand